CLINICAL TRIAL: NCT03009162
Title: A Phase I, Multicenter, Open-Label, Parallel-Group Adaptive Pharmacokinetic Single Dose Study of Oral Lasmiditan in Subjects With Normal and Impaired Renal Function
Brief Title: Study of Oral Lasmiditan in Participants With Normal and Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: CoLucid Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16895; CUD-P4-001 (Other: Algorithme Pharma); COl MIG-113 (Other: CoLucid Pharmaceuticals); H8H-CD-LAHN (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2018-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — lasmiditan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Renal impaired participants (Experimental): Participants received single 200 milligrams (mg) oral tablet of lasmiditan.
  Interventions: Drug: Lasmiditan
- Healthy participants (Experimental): Participants received single 200 mg oral tablet of lasmiditan.
  Interventions: Drug: Lasmiditan

INTERVENTIONS:
Drug: Lasmiditan — 200 mg, single oral tablet
  Other Names: LY573144

SUMMARY:
This is a multi-center, open-label, non-randomized, parallel-group, adaptive, single dose study.

This study will enroll up to 32 participants using an adaptive design that can include up to 3 groups of 8 participants with different degree of renal impairment and one group of 8 control participants with normal renal function.

Screening data will be reviewed to determine participant eligibility. Participants who meet all inclusion criteria and none of the exclusion criteria will be entered in the study.

First, approximately 16 participants will be enrolled with severe renal impairment and matched participants with normal renal function. There will be 8 participants in each of the following groups based on renal function at screening:

* Group 1: Healthy participants with normal renal function (estimated glomerular filtration rate [eGFR] ≥ 90 milliliters per minute per 1.73 meters squared [mL/min/1.73m²])
* Group 2: Severe renal impairment participants (eGFR < 30 mL/min/1.73m²) Based on safety and pharmacokinetic (PK) results from participants with severe renal impairment (Group 2), Group 3 (Moderate Renal Impairment) and Group 4 (Mild Renal Impairment) will be enrolled if substantial change in the exposure of lasmiditan is observed in participants with severe renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Motivated participant and absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements; ability to cooperate adequately; ability to understand and observe the instructions of the physician or designee
* Male or female participant
* A female participant if of childbearing potential - must be willing to use accepted contraceptive regimens from at least 28 days prior to the drug administration, during the study and for at least 60 days after the dose.
* A male participant with sexual partners who are of child bearing potential must be willing to use accepted contraceptive regimens.
* A male participant agrees to refrain from sperm donation from drug administration until 3 months after the drug administration
* Participant aged of at least 18 years
* Participant with a body mass index (BMI) ≥18.50 kilogram per meter squared (kg/m²) and < 42.00 kg/m²
* Light-, non- or ex-smokers. A light smoker is defined as someone smoking 10 cigarettes or less per day for at least 3 months before Day 1 of this study. An ex smoker is defined as someone who completely stopped smoking for at least 6 months before Day 1 of this study
* Willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the participant

Participants with Normal Renal Function:

* Clinical laboratory values within the laboratory's stated normal range; if not within this range, these must be without any clinical significance
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations (hematology, general biochemistry, electrocardiogram [ECG], and urinalysis)
* For each gender, have to match by age (± 10 years) and weight (± 20%) to the pooled mean values of participants with severe renal impairment
* Have an eGFR ≥ 90 mL/min/1.73m² calculated using Modification of Diet in Renal Disease (MDRD) equation at screening

Renal Impaired Participants:

* Considered clinically stable in the opinion of the Investigator
* Presence of mild renal impairment (eGFR 60-89 mL/min/1.73m²), moderate renal impairment (eGFR 30-59 mL/min/1.73m²), or severe renal impairment (eGFR < 30 mL/min/1.73m²) calculated using MDRD equation at screening

Exclusion Criteria:

All Participants:

* Females who are pregnant or are lactating
* History of significant hypersensitivity to lasmiditan or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases
* Participant is at imminent risk of suicide (positive response to question 4 or 5 on the Columbia-Suicide Severity Rating Scale [C-SSRS]) or had a suicide attempt within 6 months prior to screening
* Presence or history of any disorder (including Parkinson disease) that could interfere with completion of the study based on the opinion of the Principal Investigator
* Any history of tuberculosis and/or prophylaxis for tuberculosis
* Positive results to human immunodeficiency virus antigen/antibody (HIV Ag/Ab) Combo, Hepatitis B surface antigen (HBsAG (B) (hepatitis B) or Hepatitis C Virus (HCV [C]) tests
* Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 28 days before Day 1 of this study
* Females who are pregnant according to a positive pregnancy test
* Participants who took lasmiditan in the previous 28 days before Day 1 of this study
* Participants who took an Investigational Product (in another clinical trial) in the previous 28 days before Day 1 of this study
* Participants who have already participated in this clinical study
* Participants who donated 50 mL or more of blood in the previous 28 days before Day 1 of this study
* Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before Day 1 of this study

Participants with Normal Renal Function:

* Seated pulse rate less than or equal 40 Beats per Minute (bpm) or more than - Seated blood pressure below 90/60 millimeters of mercury (mmHg) or higher than 140/90 mmHg at screening
* Presence of significant gastrointestinal, liver, or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs or known to potentiate or predispose to undesired effects
* History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability, including but not limited to cholecystectomy
* Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
* Presence of out-of-range cardiac interval (PR < 110 milliseconds [msec], PR > 220 msec, QRS < 60 msec, QRS >119 msec and correct QT interval (QTc) > 450 msec for males and > 460 msec for females) on the screening ECG or other clinically significant ECG abnormalities
* Positive screening of alcohol and/or drugs of abuse
* Any clinically significant illness in the previous 28 days before Day 1 of this study

Renal Impaired Participants:

* Seated pulse rate less than 50 bpm or more than 110 bpm at screening
* Seated blood pressure below 90/50 mmHg or higher than 180/110 mmHg at screening
* Currently undergoing any method of dialysis
* History of renal transplant
* History or presence, in the opinion of the Investigator, of significant clinically unstable respiratory, cardiovascular, pulmonary, hepatic, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease,
* Have poorly controlled Type 1 or Type 2 diabetes as defined by Hemoglobin A1c >10%
* Require immunosuppressive medications for treatment of immune-mediated renal disease or kidney transplant recipients
* Evidence of renal carcinoma present at the time of screening
* Have relevant clinical laboratory abnormalities, including any elevation of alanine aminotransferase (ALT), aspartate aminotransferase (AST), or bilirubin at screening. If the investigator concludes that there is no safety risk for participants with isolated laboratory abnormalities (eg, those that do not reflect end-organ dysfunction; for example, elevated bilirubin in Gilbert's participants) to participate in the study, such cases need to be discussed and approved by the sponsor's medical monitor prior to study enrollment
* Presence of clinically significant physical, laboratory, or ECG finding that, in the opinion of the Investigator and/or sponsor, may interfere with any aspect of study conduct or interpretation of results
* Participants with acute, unstable, or untreated significant medical conditions. Participants requiring treatment for renal impairment or other chronic disease (eg, well-controlled diabetes, hypertension) must be on a stable treatment plan (medicines, doses, and regimens) for at least 2 weeks (except insulin) prior to Day 1 and during the entire study. Small adjustments in the dosages of some concomitant medications may be permitted during the study, and will be discussed on a case-by-case basis. In all cases, the participants' treatment history must be reviewed and their enrollment must be agreed to by both the investigator and the sponsor's medical monitor
* Positive screening of alcohol and/or drugs of abuse unless results can be explained by a prescription medication
* Concurrent use of medications known to affect the elimination of serum creatinine (eg, trimethoprim/sulfamethoxazole [Bactrim®] or cimetidine [Tagamet®]) and competitors of renal tubular secretion (eg, probenecid) within 30 days prior to the first dose of study drug or anticipated need for these therapies through the last pharmacokinetic (PK) sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Canada (2):
  - CIUSSS de l'est-de-l'île-de-Montréal - installation Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Algorithme Pharma, Mount Royal, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Participants: Participants received single 200 milligrams (mg) oral dose of lasmiditan.
- Renal Impaired Participants: Participants received single 200 mg oral dose of lasmiditan.
Period: Overall Study
Arm/Group | Healthy Participants | Renal Impaired Participants
Started | 8 | 8
Received at Least 1 Dose of Study Drug | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | Renal Impaired Participants | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.4 (12.3) | 51.8 (15.6) | 48.6 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 4 | 7 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax)
Description: Maximum observed plasma concentration of lasmiditan.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 36 hours, postdose
Population: All enrolled participants who received at least one dose of study drug and have evaluable pharmacokinetics (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Healthy Participants; Renal Impaired Participants: Participants received single 200 mg oral dose of lasmiditan.
Arm/Group | Healthy Participants | Renal Impaired Participants
Number analyzed (Participants) | 8 | 8
nanogram per milliliter (ng/mL) | 259 (44) | 293 (35)

2. Primary Outcome: Pharmacokinetics: Time of Maximum Observed Plasma Concentration (Tmax)
Description: Time of maximum observed plasma concentration; if it occurs at more than one time point, Tmax is defined as the first time point with this value
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 36 hours, postdose
Population: All enrolled participants who received at least one dose of study drug and have evaluable PK data.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Healthy Participants | Renal Impaired Participants
Number analyzed (Participants) | 8 | 8
hours (h) | 2.50 [1.00 to 3.00] | 1.78 [0.75 to 3.00]

3. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Zero to Tlast (AUC[0-tlast])
Description: Area Under the Concentration Versus Time Curve (AUC) from time zero to tlast (AUC[0- tlast]) of lasmiditan.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 36 hours, postdose
Population: All enrolled participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Healthy Participants | Renal Impaired Participants
Number analyzed (Participants) | 8 | 8
nanogram*hour per milliliter (ng*h/mL) | 1580 (44) | 1870 (32)

4. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-inf])
Description: Area Under the Concentration Versus Time Curve (AUC) from time zero to infinity (AUC[0-inf]) of lasmiditan.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 36 hours, postdose
Population: All enrolled participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Healthy Participants | Renal Impaired Participants
Number analyzed (Participants) | 8 | 8
ng*h/mL | 1600 (44) | 1890 (32)

5. Primary Outcome: Pharmacokinetics: Amount Excreted in Urine as Unchanged Drug or Metabolite (Ae [0-t])
Description: Amount excreted in urine (calculated as total lasmiditan concentration multiplied by volume of urine)
Time Frame: Predose and intervals: 0 to 2, 2 to 4, 4 to 8, 8 to 12, 12 to 24 and 24 to 36 hours, postdose
Population: All enrolled participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams (mg)
Arm/Group | Healthy Participants | Renal Impaired Participants
Number analyzed (Participants) | 8 | 8
milligrams (mg) | 4.64 (36) | 1.85 (45)

6. Primary Outcome: Pharmacokinetics: Fraction of Dose Excreted in Urine (fe)
Description: Fraction of dose excreted in urine (Ae / dose)
Time Frame: Predose and intervals: 0 to 2, 2 to 4, 4 to 8, 8 to 12, 12 to 24 and 24 to 36 hours, postdose
Population: All enrolled participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Healthy Participants | Renal Impaired Participants
Number analyzed (Participants) | 8 | 8
Percentage | 2.32 (36) | 0.93 (45)

7. Primary Outcome: Pharmacokinetics: Renal Clearance (CLr)
Description: Renal Clearance is the volume of blood or plasma that is completely cleared of the drug by the kidneys per unit time. (Ae(0-t)/AUC0-T)
Time Frame: Predose and intervals: 0 to 2, 2 to 4, 4 to 8, 8 to 12, 12 to 24 and 24 to 36 hours, postdose
Population: All enrolled participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour (L/h)
Arm/Group | Healthy Participants | Renal Impaired Participants
Number analyzed (Participants) | 8 | 8
Liters/hour (L/h) | 2.93 (28) | 0.992 (42)

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Safety was assessed from time of consent through end of study (up to 7 days). Data presented are the number of participants who experienced 1 or more AEs (all causalities and drug-related) and serious AEs (SAEs). A summary of SAEs and other non-serious AEs, regardless of causality is located in the Reported Adverse Events section of this record.
Time Frame: Up To 7 days
Population: All enrolled participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants | Renal Impaired Participants
Number analyzed (Participants) | 8 | 8
Participants
  Other AEs | 6 | 6
  SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Up To 7 days
Description: All enrolled participants who received at least one dose of study drug.
Arm/Group | Healthy Participants | Renal Impaired Participants
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/8 | 6/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants (N=8) | Renal Impaired Participants (N=8)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0)
Vessel puncture site erythema (General disorders) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural anxiety (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 3 (3) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the Study and its results shall not be publicized in any form without prior consent of the Sponsor. Such approval is necessary to prevent premature disclosure of trade secrets and other confidential information.

DOCUMENTS (2):
  • Study Protocol (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT03009162/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT03009162/SAP_001.pdf